CLINICAL TRIAL: NCT00438386
Title: Aripiprazole for the Treatment of Refractory Anxiety: Impact on Clinical Outcomes, Resilience and Neuroendocrinologic Parameters
Brief Title: Aripiprazole for the Treatment of Refractory Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Mark H Pollack, M.D., Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-P-000935
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Generalized Anxiety Disorder; Panic Disorder
Keywords: Generalized Anxiety Disorder; Panic Disorder; Anxiety Disorder; Aripiprazole
MeSH Terms: conditions — Generalized Anxiety Disorder; Panic Disorder; Anxiety Disorders | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The purpose of this study is to determine whether aripiprazole is effective in the treatment of refractory panic and generalized anxiety disorder.

DETAILED DESCRIPTION:
Accruing evidence demonstrates that the anxiety disorders are common and associated with significant morbidity and impairment. Although current first-line interventions are effective, many patients remain at least somewhat symptomatic, and some respond not at all, despite initial treatment. For instance, Generalized Anxiety Disorder (GAD) is a common distressing and disabling condition affecting 5% of the population. It is typically characterized by a chronic course and associated with significant psychosocial impairment and decreased quality of life (Simon and Pollack 2000). Although a number of therapeutic agents have demonstrated efficacy in the treatment of GAD, only a minority of anxious patients experience remission with initial treatment.

Panic disorder with or without agoraphobia is a common anxiety disorder, occurring in 3.5 % of the population (Kessler, et al., 1994). Although the study of panic disorder has advanced in recent years, with the availability of a growing number of treatments with reported efficacy in clinical trials and practice, acute and longitudinal follow-up studies of patients with panic disorder suggest that many individuals remain symptomatic despite treatment (Pollack and Otto, 1994). However, there is no systematic data currently available to guide the treatment of patients with panic disorder who remain symptomatic after initial intervention.

Thus, one purpose of this study is to examine the efficacy of the addition of aripiprazole, for the treatment of patients with GAD or panic disorder who remain refractory despite a treatment trial with an anxiolytic (e.g. antidepressant, benzodiazepine, buspirone). Aripiprazole is a novel antipsychotic agent with potent effects at the serotonergic, as well as dopaminergic receptor, and a more favorable side effect profile than standard neuroleptics, including a low potential to cause extrapyramidal symptoms.

The study period is a 9-week, acute treatment phase. Patients who meet inclusion criteria will receive aripiprazole for 8 weeks. Treatment will be initiated with 2.5 mg/day at the baseline visit, 5 mg/day aripiprazole for the first week and flexibly titrated up to a maximum of 30 mg/day over the next six weeks. Patients will be seen weekly for the first three weeks of this phase of treatment, and then at 2-week intervals for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, age 18-75.
* Diagnosis of Generalized Anxiety Disorder (GAD) or Panic Disorder (PD) with or without Agoraphobia.
* For GAD: Hamilton Anxiety Rating Scale score greater than or equal to 16, and for PD: MGH Anchored Panic CGI Severity Rating greater than or equal to 4.
* Hamilton Depression Scale score less than or equal to 18.5) Clinical Global Impression of Severity score Score equal to or greater than 4.
* History of persistent anxiety despite at least 8 weeks of an adequate (or highest tolerated) dose of anxiolytic pharmacotherapy. This is operationalized to include an antidepressant (e.g., paroxetine 20 mg/d; imipramine 150 mg/d or phenelzine 60 mg/d or their equivalent) or a benzodiazepine (e.g., clonazepam 2 mg/d or its equivalent). The dose of medication should be stable for at least 2 weeks prior to evaluation.
* Willingness and ability to comply with the requirements of the study protocol.

Exclusion Criteria:

* Pregnant or lactating women or others not using acceptable means of birth control (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, implanted progesterone rods stabilized for at least 3 months).
* Patients with current or history of bipolar disorder, schizophrenia or other psychotic conditions.
* Patients with a history of alcohol or substance abuse or dependence within the last six months or a positive toxicology screen for drugs of abuse at baseline.
* Patients with significant unstable medical illness or illness which results in HPA axis dysregulation, or other neurohormonal dysregulation.
* Severe personality disorders likely to interfere with study participation.
* Ongoing psychotherapy directed toward the treatment of the primary anxiety disorder.
* History of hypersensitivity to aripiprazole, or > 1 previous treatment failure for anxiety with atypical antipsychotics. Concomitant treatment with other antipsychotics
* Patients exhibiting suicidality as evidenced by a score greater than 2 on item #3 of the HAM-D.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale
Clinician Global Impression-Severity
Connor Davidson Resilience Scale

SECONDARY OUTCOMES:
Panic Disorder Severity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Pollack, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Anxiety and Traumatic Stress Disorders at Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Simon NM, Pollack MH. The Current Status of the Treatment of Panic Disorder: Pharmacotherapy and Cognitive-Behavioral Therapy. Psych Ann 30(11): 689-696, 2000.
- [Background] Kessler RC, McGonagle KA, Zhao S, Nelson CB, Hughes M, Eshleman S, Wittchen HU, Kendler KS. Lifetime and 12-month prevalence of DSM-III-R psychiatric disorders in the United States. Results from the National Comorbidity Survey. Arch Gen Psychiatry. 1994 Jan;51(1):8-19. doi: 10.1001/archpsyc.1994.03950010008002. PMID 8279933
- [Background] Pollack, M, Otto, M. Long-Term Pharmacologic Treatment of Panic Disorder. Psychiatric Annals 24: 291-298, 1994.